CLINICAL TRIAL: NCT03918850
Title: Medication Treatment for Opioid Use Disorder in Expectant Mothers (MOMs): a Pragmatic Randomized Trial Comparing Extended-release and Daily Buprenorphine Formulations
Brief Title: Medication Treatment for Opioid Use Disorder in Expectant Mothers
Acronym: MOMs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: T. John Winhusen, PhD (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor-Investigator, T. John Winhusen, PhD, Professor; Vice Chair and Division Director of Addiction Sciences, University of Cincinnati
Organization: University of Cincinnati (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0429-1; UG1DA013732 (NIH)
Record Dates: First submitted 2019-04-09; First posted 2019-04-18 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Opioid-Related Disorders; Drug Addiction; Pregnancy Related; Substance Abuse; Drug Abuse; Neonatal Abstinence Syndrome; Neonatal Opioid Withdrawal Syndrome; Drug Abuse in Pregnancy
Keywords: CTN-0080; clinical trials network; medication assisted treatment
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders; Neonatal Abstinence Syndrome | interventions — Buprenorphine; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Intervention Model Description: This is an intent-to-treat, two-arm, open-label, pragmatic randomized controlled trial.
Masking Description: The primary outcome is assessed in a masked fashion by a central laboratory, but there is no masking for other outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BUP-XR (Experimental): Weekly subcutaneous Buprenorphine Injection (CAM2038) during pregnancy. During the 12-month postpartum phase, participants who are breastfeeding will continue receiving subcutaneous Buprenorphine Injection weekly; participants who are not breastfeeding will receive subcutaneous Buprenorphine Injection monthly.
  The target doses will be 24 mg for the weekly formulation and 96 mg for the monthly formulation, but the actual dose may be lower or higher as determined by the prescribing clinician (e.g., based on craving/withdrawal experienced by the participant, etc.).
  Interventions: Drug: Buprenorphine Injection
- BUP-SL (Active Comparator): Daily sublingual buprenorphine, with or without naloxone, based on site preference, during pregnancy and during the 12-month postpartum phase.
  The target dose will be 16 mg daily, but the actual dose may be lower or higher as determined by the prescribing clinician (e.g., based on craving/withdrawal experienced by the participant, etc.).
  Interventions: Drug: Buprenorphine Sublingual Product

INTERVENTIONS:
Drug: Buprenorphine Injection — Weekly and monthly formulations of injectable, extended-release buprenorphine (BUP-XR).
  Other Names: CAM2038
  Arms: BUP-XR
Drug: Buprenorphine Sublingual Product — Sublingual buprenorphine (BUP-SL), administered daily.
  Other Names: Subutex; Suboxone
  Arms: BUP-SL

SUMMARY:
The primary objective of this study is to evaluate the impact of treating opioid use disorder (OUD) in pregnant women with extended-release buprenorphine (BUP-XR), compared to sublingual buprenorphine (BUP-SL), on mother and infant outcomes. The primary hypothesis is that the BUP-XR group will not have greater illicit opioid use than the BUP-SL group during pregnancy (non-inferiority).

DETAILED DESCRIPTION:
This is an intent-to-treat, two-arm, open-label, pragmatic randomized controlled trial. Eligible participants will be randomized in a 1:1 ratio to BUP-XR or BUP-SL, balancing on site, estimated gestational age (EGA) at time of randomization (6 weeks-18 weeks vs. 19 weeks-30 weeks), and whether they are on BUP-SL at the time of randomization (yes vs. no). Participants will be provided with study medication and attend weekly medication visits through 12 months postpartum.

ELIGIBILITY:
Inclusion Criteria:

Potential participants must:

1. be 18-41 years of age
2. be pregnant with an estimated gestational age (EGA) of 6 - 30 weeks at randomization, has evidence of a viable intrauterine pregnancy if EGA < 12 weeks and is not planning to terminate the pregnancy
3. have a single fetus pregnancy (can be based on self-report if an objective assessment is unavailable)
4. meet Diagnostic and Statistical Manual (DSM)-5 criteria for moderate/severe OUD and be a good candidate for BUP maintenance and/or be currently prescribed BUP for the treatment of OUD
5. be willing to be randomized to BUP-XR or BUP-SL and to comply with study procedures, including weekly Medication Check Visits
6. be planning to deliver at one of the hospitals for which the BORN survey was completed and that: a) has a written protocol for the management of neonatal abstinence syndrome (NAS) / neonatal withdrawal syndrome (NOWS), b) offers rooming-in while infants are being observed for NAS/NOWS; and c) does not send infants home on opioids for the treatment of NAS/NOWS
7. be enrolled in outpatient addiction treatment at a participating site (e.g., have completed intake)
8. be able to understand the study, and having understood, provide written informed consent in English

Exclusion Criteria:

Potential participants must not:

1. have a physiological dependence on alcohol or sedatives requiring medical detoxification
2. have a psychiatric condition that, in the judgment of the site medical clinician (MC), would make study participation unsafe or which would make treatment compliance difficult. Examples include:

   * Suicidal or homicidal ideation requiring immediate attention
   * Severe, inadequately-treated mental health disorder (e.g., active psychosis, uncontrolled bipolar disorder)
3. have a medical condition that, in the judgment of the study MC, would make study participation unsafe or which would make treatment compliance difficult. Medical conditions that may compromise participant safety or study conduct include, but are not limited to, allergy/sensitivity to study medications and the following based on clinical labs:

   * aspartate aminotransferase (AST) / alanine aminotransferase (ALT) greater than 5X upper limit of normal
   * serum creatinine greater than 1.5X upper limit of normal
   * total bilirubin greater than 1.5X upper limit of normal
4. be currently in jail, prison or any inpatient overnight facility as required by court of law or have pending legal action or other situation (e.g., unstable living arrangements) that, in the judgement of the site investigator, could prevent participation in the study or in any study activities;
5. be currently receiving methadone or naltrexone for the treatment of OUD;
6. be enrolled in or planning to enroll in treatment beyond the level 3.3 (Clinically Managed Population-Specific High-Intensity Residential Services) of the American Society of Addiction Medicine criteria; for level 3.3, the participant must have the ability to leave the facility unaccompanied by staff as needed;
7. be enrolled in or planning to enroll in: a) a trial testing medication for managing OUD during pregnancy; b) research testing an intervention for substance use disorder or NOWS in their infant unless they are willing to provide a release for the research records.

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Proportion of illicit opioid-negative urine samples during pregnancy | Screening through delivery
  Weekly urine samples are shipped to a central laboratory, where they are analyzed for presence of illicit opioids and/or their metabolites.

SECONDARY OUTCOMES:
Total days of neonatal opioid treatment during the hospital stay | Neonate discharge from hospital, typically within 1 month postpartum
  This outcome will be abstracted from the medical record.
Proportion of illicit opioid-negative urine samples postpartum | Delivery through 12 months postpartum
  Weekly urine samples are shipped to a central laboratory, where they are analyzed for presence of illicit opioids and/or their metabolites.
Proportion of days with study medication adherence | Screening through 12 months postpartum
  Adherence to treatment during pregnancy through 12 months postpartum
Proportion of drug and alcohol-negative urine samples | Screening through 12 months postpartum
  Weekly urine samples are shipped to a central laboratory, where they are analyzed for presence of alcohol, illicit drugs and/or their metabolites.
Opioid Craving Scale | Screening through delivery
  The scale consists of 3 items, measuring craving, cue-induced craving, and likelihood of using, rated on a visual analogue scale from 0-10. The total is calculated by averaging the 3 item scores. Higher scores indicate greater levels of opioid craving.
Opioid Craving Scale | Delivery through 12 months postpartum
  The scale consists of 3 items, measuring craving, cue-induced craving, and likelihood of using, rated on a visual analogue scale from 0-10. The total is calculated by averaging the 3 item scores. Higher scores indicate greater levels of opioid craving.
Adequacy of Prenatal Care Utilization Index | At delivery
  The information will be derived from either medical records or the birth certificate.
Short Opiate Withdrawal Scale (SOWS)-Gossop | Screening through 12 months postpartum
  Measure of maternal opioid withdrawal symptoms.
Opioid Medication for Neonatal Opioid Withdrawal Syndrome (NOWS) Symptoms | Neonate discharge from hospital, typically within 1 month postpartum
  Use of opioid medication for NOWS symptoms will be abstracted from the medical record.
Infant Hospital Length of Stay | Neonate discharge from hospital, typically within 1 month postpartum
  Infant hospital length of stay (LOS) defined as the infant's age, in days, at discharge will be abstracted from the medical record. (Infant)
Adjunct Medications | Neonate discharge from hospital, typically within 1 month postpartum
  Use of adjunct medications (e.g., phenobarbital, clonidine) will be abstracted from the medical record.
Neonatal Opioid Withdrawal Syndrome (NOWS) Peak Score | Neonate discharge from hospital, typically within 1 month postpartum
  NOWS peak score will be abstracted from the medical record. Because sites may use different NOWS scoring systems, the scoring system that was used will be included as part of the peak score abstraction.
Diagnosis code for Neonatal Opioid Withdrawal Syndrome (NOWS) | Neonate discharge from hospital, typically within 1 month postpartum
  A diagnosis code indicative of NOWS (Yes/No) will be abstracted from the medical record.
Custody at discharge | Neonate discharge from hospital, typically within 1 month postpartum
  For example, whether the infant is discharged in custody of mother, other relative, foster/adoptive family, etc. This will be abstracted from the medical record.
Medications at discharge | Neonate discharge from hospital, typically within 1 month postpartum
  Medications that the infant is to continue receiving at discharge will be abstracted from the medical record.
Child protective services open case | Neonate discharge from hospital, typically within 1 month postpartum
  Whether or not there is an open child protective services at discharge (yes/no) will be abstracted from the medical record.
Ages and Stages Questionnaire, third edition (ASQ-3) | 6 months postpartum
  To screen for developmental issues in the infant.
Ages and Stages Questionnaire, third edition (ASQ-3) | 12 months postpartum
  To screen for developmental issues in the infant.

CONTACTS AND LOCATIONS:
Overall Officials: T. John Winhusen, PhD, Principal Investigator — University of Cincinnati
Locations (12):
- United States (12):
  - Gateway Community Services, Jacksonville, Florida
  - Massachusetts General Hospital HOPE Clinic, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - University of New Mexico Milagro Clinic, Albuquerque, New Mexico
  - University of Cincinnati Health Perinatal Addictions Program, Cincinnati, Ohio
  - CODA, Inc., Portland, Oregon
  - Pregnancy Recovery Center at Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Utah SUPeRAD Clinic, Salt Lake City, Utah
  - Addiction Recovery Services (ARS), Swedish Medical Center, Seattle, Washington
  - Marshall Health MARC Program, Huntington, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
Data will be transmitted by the study Data and Statistics Center to the designated party for de-identification, posting, storing, and archiving on NIDA's Data Share website. Data Share is an online repository of data from studies funded by the National Institute on Drug Abuse. All de-identified individual participant data is expected to be made available.
Supporting Information: Study Protocol
URL: https://datashare.nida.nih.gov/

REFERENCES:
- [Derived] Krans EE, Lewis D, Douaihy A, Lofwall MR, Kropp F, Martin PR, Sanghani RS, Cottrell JN, Winhusen TJ. Cigarette use and smoking cessation goals among pregnant women with opioid use disorder. J Subst Use Addict Treat. 2025 Dec 20:209865. doi: 10.1016/j.josat.2025.209865. Online ahead of print. PMID 41429292
- [Derived] Cash E, Cochran G, Smid MC, Charles JE, Humiston G, Wei Y, Mauerman N, Carlston K, Broussard G, Sengpraseut B, Martin PR, Winhusen TJ. Overdose risk profiles in pregnancy: Latent class analysis of pregnant individuals with opioid use disorder. J Subst Use Addict Treat. 2025 Sep 25:209809. doi: 10.1016/j.josat.2025.209809. Online ahead of print. PMID 41015387
- [Derived] Winhusen TJ, Kropp F, Greenfield SF, Krans EE, Lewis D, Martin PR, Gordon AJ, Davies TH, Wachman EM, Douaihy A, Parker K, Xin X, Jalali A, Lofwall MR. Trauma Prevalence and Its Association With Health-related Quality of Life in Pregnant Persons With Opioid Use Disorder. J Addict Med. 2025 Jan-Feb 01;19(1):20-25. doi: 10.1097/ADM.0000000000001366. Epub 2024 Aug 6. PMID 39105509
- [Derived] Kropp FB, Smid MC, Lofwall MR, Wachman EM, Martin PR, Murphy SM, Wilder CM, Winhusen TJ. Collaborative care programs for pregnant and postpartum individuals with opioid use disorder: Organizational characteristics of sites participating in the NIDA CTN0080 MOMs study. J Subst Use Addict Treat. 2023 Jun;149:209030. doi: 10.1016/j.josat.2023.209030. Epub 2023 Apr 4. PMID 37023858

DOCUMENTS (1):
  • Informed Consent Form (2022-11-22): https://cdn.clinicaltrials.gov/large-docs/50/NCT03918850/ICF_000.pdf